CLINICAL TRIAL: NCT00981396
Title: The Effect of EFT (Emotional Freedom Techniques) in Smokers Failing a Smoking Cessation Program
Brief Title: The Effect of Emotional Freedom Techniques (EFT) in Smokers Failing a Smoking Cessation Program
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Investigator, Soul Medicine Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMI-SMO-92509
Record Dates: First submitted 2009-09-19; First posted 2009-09-22 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Smoking
Keywords: smoking; EFT (Emotional Freedom Techniques); CBT (cognitive behavior therapy); cravings; trauma
MeSH Terms: conditions — Smoking; Color Vision Defects; Wounds and Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: CBT (Cognitive Behavioral Therapy)
- EFT (Experimental): Emotional Freedom Techniques, a novel but efficacious stress-reduction technique
  Interventions: Behavioral: EFT (Emotional Freedom Techniques)

INTERVENTIONS:
Behavioral: EFT (Emotional Freedom Techniques) — EFT is a brief but efficacious stress-reduction intervention. It combines exposure, cognitive structuring, and somatic stimulation.
  Arms: EFT
Behavioral: CBT (Cognitive Behavioral Therapy) — CBT is a behavioral intervention that seeks to challenge and change negative client cognitions about events and life circumstances.
  Arms: CBT

SUMMARY:
The National Health Service (NHS) stop smoking service at the Central Lancashire NHS Trust serves a diverse population of smokers, with a very good quit rate and high standards. However, clinical experience predicts that some clients are unlikely to succeed through the NHS smoking cessation program. This special population has difficulty quitting for a variety of reasons. Some relapse over the course of the following two years and return repeatedly to the service. Others, for instance those with health problems, may be highly motivated to quit, but unable to resist their cravings. The purpose of this study is to determine if EFT makes a difference in quit rates with the most challenging population of clients.

ELIGIBILITY:
Inclusion Criteria:

* High anxiety related to the quit attempt
* Cravings which sabotage the quit attempt
* Low confidence at their ability to quit and remain quit

Exclusion Criteria:

* None, all NHS clients are eligible

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quit rate | treatment period

SECONDARY OUTCOMES:
Psychological symptoms and physiological symptoms | Three, 6, and 12 months after intervention
  Symptoms and smoking 3, 6 and 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- NHS Central Lancashire Primary Care Trust, Ormskirk, Lancashire, United Kingdom